CLINICAL TRIAL: NCT00837356
Title: A Multi-centre, Multi-national Open-label Sequential Trial Comparing Pharmacokinetics and Safety of N8 and Advate® in Subjects With Haemophilia A
Brief Title: Comparison of the Action of Drugs in the Body and Safety of N8 and Advate® in Haemophilia A Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN7008-3522; 2008-002157-21 (EudraCT Number)
Record Dates: First submitted 2009-02-04; First posted 2009-02-05 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Congenital Bleeding Disorder; Haemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII; recombinant factor VIII N8; recombinant FVIII, sugar formulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Advate®/turoctocog alfa (Experimental)
  Interventions: Drug: Advate®; Drug: turoctocog alfa

INTERVENTIONS:
Drug: Advate® — Subjects will receive Advate® at a dose of 50 IU/kg body weight in the first session
Drug: turoctocog alfa — After a washout period of 4 days, subjects will subsequently receive turoctocog alfa (recombinant factor VIII (N8)) at a dose of 50 IU/kg body weight in the second session
  Other Names: recombinant FVIII; N8

SUMMARY:
This trial is conducted in Europe and Asia. The aim of this clinical trial is to compare two recombinant factor VIII drugs, turoctocog alfa (recombinant factor VIII (N8)) with Advate®, in haemophilia A subjects, investigating the action and safety of the drugs.

ELIGIBILITY:
Inclusion Criteria:

* Severe haemophilia A (FVIII level less than or equal to 1%)
* Treatment history of more than 150 exposure days with recombinant or plasma-derived FVIII replacement products
* HIV or HCV negative, or if positive the patient is on a stable antiviral regimen at the time of the enrolment in the trial

Exclusion Criteria:

* Presence of any bleeding disorder in addition to haemophilia A
* Inhibitor titre greater than or equal to 0.6 Bethesda Units (BU) at screening and past history of inhibitor
* Abnormal renal function tests
* Known hypersensitivity to Advate®

Ages: 12 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2009-03; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Recovery of FVIII 30 min after administration, half-life, AUC, and clearance | at 30 days

SECONDARY OUTCOMES:
Inhibitor development | at 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (7):
- Germany (2):
  - Novo Nordisk Investigational Site, Berlin
  - Novo Nordisk Investigational Site, Hanover
- Novo Nordisk Investigational Site, Tel Litwinsky, Israel
- Italy (2):
  - Novo Nordisk Investigational Site, Florence
  - Novo Nordisk Investigational Site, Milan
- Novo Nordisk Investigational Site, Madrid, Spain
- Novo Nordisk Investigational Site, Zurich, Switzerland

REFERENCES:
- [Result] Martinowitz U, Bjerre J, Brand B, Klamroth R, Misgav M, Morfini M, Santagostino E, Tiede A, Viuff D. Bioequivalence between two serum-free recombinant factor VIII preparations (N8 and ADVATE(R))--an open-label, sequential dosing pharmacokinetic study in patients with severe haemophilia A. Haemophilia. 2011 Nov;17(6):854-9. doi: 10.1111/j.1365-2516.2011.02495.x. Epub 2011 Mar 28. PMID 21443634
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com